CLINICAL TRIAL: NCT06922097
Title: Treating Intraoperative Bradycardia in Non-cardiac Surgery Patients With Atropine at Heart Rates Below 60 Versus 30 Beats Per Minute and Norepinephrine Requirements: the Randomized RAPID Trial
Brief Title: Treating Intraoperative Bradycardia in Non-cardiac Surgery Patients With Atropine at Heart Rates Below 60 Versus 30 Beats Per Minute and Norepinephrine Requirements
Acronym: RAPID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. Alina Bergholz, MD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-101426-BO-ff
Record Dates: First submitted 2025-03-23; First posted 2025-04-10 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-04

CONDITIONS: Intraoperative Bradycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giving atropine at heart rates below 60 beats per minute (Experimental)
  Interventions: Drug: Giving atropine at heart rates below 60 beats per minute
- Giving atropine at heart rates below 30 beats per minute (Active Comparator)
  Interventions: Drug: Giving atropine at heart rates below 30 beats per minute

INTERVENTIONS:
Drug: Giving atropine at heart rates below 60 beats per minute — In patients assigned to the atropine therapy at heart rates below 60 beats per minute, atropine will be given at a dose of 0.5 mg when heart rate is below 60 beats per minute for one continuous minute. A second and third atropine dose of 0.5 mg will be given if heart rate remains or again drops below 60 beats per minute for one continuous minute. Patients will not be given more than 1.5 mg atropine.
  Arms: Giving atropine at heart rates below 60 beats per minute
Drug: Giving atropine at heart rates below 30 beats per minute — In patients assigned to atropine therapy at heart rates below 30 beats per minute, atropine will be given at a dose of 0.5 mg when heart rate is below 30 beats per minute for one continuous minute. A second and third atropine dose of 0.5 mg will be given if heart rate remains or again drops below 30 beats per minute for one continuous minute. Patients will not be given more than 1.5 mg atropine.
  Arms: Giving atropine at heart rates below 30 beats per minute

SUMMARY:
The RAPID trial is a randomized, single-center trial investigating whether giving atropine at heart rates below 60 beats per minute versus giving atropine only at heart rates below 30 beats per minute reduces the amount of norepinephrine needed to keep MAP above 65 mmHg in non-cardiac surgery patients with intraoperative bradycardia.

ELIGIBILITY:
Inclusion Criteria: Consenting patients ≥50 years scheduled for elective non-cardiac surgery with general anesthesia that is expected to last ≥60 minutes with at least two of the following risk criteria for developing acute kidney injury:

* Age ≥65 years
* American Society of Anesthesiologists physical status III or IV
* Chronic arterial hypertension
* Diabetes mellitus requiring medication
* Intraabdominal surgery
* Preoperative renal insufficiency (serum creatinine ≥1.2 mg/dL)

Exclusion Criteria:

Patients with the following exclusion criteria: contraindication for atropine administration (e.g., myasthenia gravis, high-grade aortic stenosis, high-grade coronary artery disease, glaucoma, paralytic ileus, prostatic hypertrophy); renal replacement therapy within the previous 3 months; chronic kidney disease with an estimated glomerular filtration rate <20 mL/min/1.73 m2; pregnancy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Average norepinephrine infusion rate | Perioperative
  Average norepinephrine infusion rate in μg per kg actual body weight per minute (μg kg-1 min-1) needed to keep MAP above 65 mmHg from anesthetic induction until the end of surgery (continuous outcome)

SECONDARY OUTCOMES:
Time-weighted average MAP <65 mmHg | Perioperative
  From anesthetic induction until the end of surgery
Time-weighted average heart rate <60 bpm | Perioperative
  From anesthetic induction until the end of surgery
Time-weighted average MAP >110 mmHg | Perioperative
  From anesthetic induction until the end of surgery
Time-weighted average heart rate >100 bpm | Perioperative
  From anesthetic induction until the end of surgery

OTHER OUTCOMES:
Incidence of acute kidney injury | Within the first 3 postoperative days
  Acute kidney injury (binary outcome) will be defined as an increase in postoperative creatinine of ≥50 % from baseline.
Incidence of delirium | Within the first 3 postoperative days
  Delirium (binary outcome) will be assessed twice daily within the first three postoperative days using the 3-Minute Diagnostic Confusion Assessment Method for patients on normal wards and the Confusion Assessment Method for Intensive Care Unit for patients in intensive care units.
Incidence of urinary retention | Within the first 3 postoperative days
  Urinary retention (binary outcome) will be assessed by reviewing the diagnoses documented in the patients' medical records within the first 3 postoperative days.
Incidence of central anticholinergic syndrome | Within the first 3 postoperative days
  Central anticholinergic syndrome (binary outcome) will be assessed by reviewing the diagnoses documented in the patients' medical records within the first 3 postoperative days.
Incidence of acute angle-closure glaucoma | Within the first 3 postoperative days
  Acute angle-closure glaucoma (binary outcome) will be assessed by reviewing the diagnoses documented in the patients' medical records within the first 3 postoperative days.

CONTACTS AND LOCATIONS:
Overall Officials: Alina Bergholz, MD, Principal Investigator — University Medical Centre Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No